CLINICAL TRIAL: NCT04052776
Title: Acute Effects of Pharmacological Neuromodulation on Leg Motor Activity in Patients With Spinal Cord Injury Treated With Epidural Electrical Stimulation
Brief Title: Acute Effects of Pharmacological Neuromodulation on Leg Motor Activity in Patients With SCI Treated With EES
Acronym: STIMO-PHARMA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, Jocelyne Bloch, Professor Medical Doctor, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-01057
Record Dates: First submitted 2019-07-29; First posted 2019-08-12 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Spinal Cord Injuries; Drug Effect
Keywords: Pharmacology; Neuromodulation; Epidural electrical stimulation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Buspirone; carbidopa, levodopa drug combination

STUDY DESIGN:
Intervention Model Description: This study will be monocentric, randomized, double-blind, placebo-controlled with a four-sequence crossover design.
  All participants will undergo the 4 treatment arms. and each of them will be their own control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded and undistinguishable pills will be made by a pharmacy laboratory in order to conceal their nature from the clinicians and the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Buspirone (Active Comparator): 40mg
  Interventions: Drug: Buspirone
- Levodopa-Carbidopa (Active Comparator): 400mg/100mg
  Interventions: Drug: Levodopa-Carbidopa
- Buspirone + Levodopa-Carbidopa (Active Comparator): 40mg + 400mg/100mg
  Interventions: Drug: Buspirone + Levodopa-Carbidopa
- Placebo (Placebo Comparator): Mannitol pill
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Buspirone — 40mg
  Arms: Buspirone
Drug: Levodopa-Carbidopa — 400mg/100mg
  Arms: Levodopa-Carbidopa
Drug: Buspirone + Levodopa-Carbidopa — 40mg + 400mg/100mg
  Arms: Buspirone + Levodopa-Carbidopa
Drug: Placebo oral tablet — Non-active metabolite
  Arms: Placebo

SUMMARY:
In a current first-in-man study, called Stimulation Movement Overground (STIMO) (NCT02936453; CER-VD: 04-2014; Swissmedic: 2016-MD-0002), epidural electrical stimulation (EES) of the spinal cord is applied to enable individuals with severe spinal cord injury (SCI) to complete intensive locomotor neurorehabilitation training. In this clinical feasibility study, it was demonstrated that EES results in an immediate enhancement of locomotor functions and that when applied repeatedly as part of a neurorehabilitation program, EES can progressively improve leg motor control in individuals with severe SCI. Mechanistically, EES acts trans-synaptically upon spinal circuitries through the electrical stimulation of proprioceptive fibers.

It is assumed that this stimulation does not increase the level of availability of monoamine neurotransmitters below the SCI level, which are essential for lower extremity movement generation. Specifically, in a non-injured individual, dopamine and serotonin synthesized in the brain and brainstem are released by fibers diffusely innervating the spinal cord, serving to critically mediate excitability of motor neurons and interneurons in lumbar and sacral spinal level. Spinal cord injury would partially or entirely disrupt these modulation pathways, resulting in a detrimental lack of crucial neurotransmitters below the injury level. This lack of endogenous neurotransmitters could potentially be compensated for by pharmacological agents promoting the neurochemical environment necessary for locomotion.

DETAILED DESCRIPTION:
The aim is to test the effects of orally administered buspirone and levodopa/carbidopa taken individually and in combination. Both buspirone and levodopa can cross the blood-brain barrier, and reach the lumbar spinal cord where 5-HT1A receptors are expressed, and levodopa can presumably be synthesized by specialized dopaminergic into dopamine. Alternatively, levodopa effects might be mediated via noradrenaline, following dopamine metabolization. Therefore, it is hypothesized that the combination of pharmacological neuromodulation with EES would further improve locomotor functions and lower extremity motor score.

The primary and safety objective is to evaluate the safety and the tolerability of a single-dose of immediate-release levodopa/carbidopa, buspirone, the combination levodopa/carbidopa and buspirone, and the placebo in individuals with SCI.

The secondary objectives are to assess the following effects of levodopa/carbidopa, buspirone, the combination levodopa/carbidopa and buspirone, and the placebo on the lower extremities:

1. Spasticity
2. Lower Extremity Motor score (LEMS)
3. Voluntary movements
4. Gait patterns and velocity Participants' safety will be ensured with the usage of Rysen, which a CE-marked bodyweight support system robot, and the aid of locomotor assistive device.

ELIGIBILITY:
Inclusion Criteria:

* Completed the main phase of the STIMO study
* Enrolled in the STIMO study extension
* Age 18-65 (women or men)
* Sensorimotor or motor complete and incomplete SCI graded as AIS A, B, C & D
* Stable medical, physical and psychological condition as considered by Investigators
* Able to understand and interact with the study team in French or English
* Adequate caregiver support and access to appropriate medical care in the patient's home community
* Agree to comply with all conditions of the study and to attend all required study training and visit
* Must provide and sign Informed Consent prior to any study-related procedures

Exclusion Criteria:

* Epilepsy
* Women who are pregnant (pregnancy test obligatory for women of childbearing potential) or breastfeeding or not willing to take contraception.
* Known or suspected non-compliance, drug or alcohol abuse.
* Gastrointestinal ulcers in the last five years
* Known or suspected eye disorders or diseases
* Known or suspected allergies or hypersensitivity to buspirone, levodopa or carbidopa.
* Taking selective and non-selective serotonin reuptake inhibitors or any other treatments acting upon serotonergic transmission, such as the following:

  * Selective serotonin reuptake inhibitors (SSRIs)
  * Serotonin-norepinephrine reuptake inhibitors (SNRIs)
  * Serotonin antagonists and reuptake inhibitors (SARIs)
  * Tricyclic antidepressants (TCAs)
  * Tetracyclic antidepressants (TeCAs)
  * Norepinephrine-dopamine reuptake inhibitors (NDRIs)
  * Monoamine oxidase inhibitors (MAOIs)
* Patients who are receiving treatments altering the noradrenergic and dopaminergic transmission (e.g., bupropion and levodopa/carbidopa)
* Patients who are taking narcotic pain killers (e.g., opioids) and neuropathic medication (e.g., gabapentin, pregabalin)
* Patients who are taking antihypertensive drugs and diuretics (e.g., furosemide or hydrochlorothiazide)
* Patients who are taking hypnotic drugs (e.g., Zolpidem).
* Patients receiving D2 antagonists or antipsychotic drugs (e.g., butyrophenone, phenothiazines, risperidone)
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Rate of AEs/SAEs/Side effects | Changes from baseline condition over a treatment session of 4 hours
  Evaluate the safety of oral, single-dose administration of levodopa/carbidopa, buspirone, the combination of buspirone and levodopa/carbidopa, and placebo.
  * The frequency and the severity AEs and SAEs will be collected thoughout the treatment session
  * Reported side effects throughout the treatment sessions will also be collected by a tailored quantitative/qualitative questionnaire
Changes in blood pressure | Changes from baseline condition over a treatment session of 4 hours
  Evaluate the safety of oral, single-dose administration of levodopa/carbidopa, buspirone, the combination of buspirone and levodopa/carbidopa, and placebo
  -Vitals signs will be monitored throughout the treatment session to evaluate the fluctuations from baseline condition.
Changes in heart rate | Changes from baseline condition over a treatment session of 4 hours
  Evaluate the safety of oral, single-dose administration of levodopa/carbidopa, buspirone, the combination of buspirone and levodopa/carbidopa, and placebo
  -Vitals signs will be monitored throughout the treatment session to evaluate the fluctuations from baseline condition.

SECONDARY OUTCOMES:
Spasticity of the Lower Extremities (score according to the Pendulum test) | Changes from baseline condition over a treatment session of 4 hours
  Explore preliminary efficacy of oral, single-dose administration of levodopa/carbidopa, buspirone, the combination of buspirone and levodopa/carbidopa, and placebo.
  -Assessment of the lower extremities' spasticity.
Lower Extremity Motor Strength (M0-M5 score according to the AIS) | Changes from baseline condition over a treatment session of 4 hours
  Explore preliminary efficacy of oral, single-dose administration of levodopa/carbidopa, buspirone, the combination of buspirone and levodopa/carbidopa, and placebo.
  -Assessment of the lower extremities' motor strength by a clinician.
Lower Extremity Motor Strength (muscle activity) | Changes from baseline condition over a treatment session of 4 hours
  Explore preliminary efficacy of oral, single-dose administration of levodopa/carbidopa, buspirone, the combination of buspirone and levodopa/carbidopa, and placebo.
  -Assessment of the lower extremities' motor strength by EMGs.
Lower Extremity Voluntary Movements (kinematics assessment through VICON) | Changes from baseline condition over a treatment session of 4 hours
  Explore preliminary efficacy of oral, single-dose administration of levodopa/carbidopa, buspirone, the combination of buspirone and levodopa/carbidopa, and placebo.
  -Participants' voluntary movements will be assessed by kinematics analyses through the VICON)
Lower Extremity Voluntary Movements (muscle activity) | Changes from baseline condition over a treatment session of 4 hours
  Explore preliminary efficacy of oral, single-dose administration of levodopa/carbidopa, buspirone, the combination of buspirone and levodopa/carbidopa, and placebo.
  -Participants' muscles during the voluntary movements will be assessed by EMGs.
Walking speed (10MWT) | Changes from baseline condition over a treatment session of 4 hours
  Explore preliminary efficacy of oral, single-dose administration of levodopa/carbidopa, buspirone, the combination of buspirone and levodopa/carbidopa, and placebo.
  -Participants' velocity will be assessed with a 10MWT with and without EES
Gait pattern (kinematics assessment through VICON) | Changes from baseline condition over a treatment session of 4 hours
  Explore preliminary efficacy of oral, single-dose administration of levodopa/carbidopa, buspirone, the combination of buspirone and levodopa/carbidopa, and placebo.
  -Participants' gait pattern during a 10MWT will be assessed by kinematics analyses through the VICON
Gait pattern (muscle activity) | Changes from baseline condition over a treatment session of 4 hours
  Explore preliminary efficacy of oral, single-dose administration of levodopa/carbidopa, buspirone, the combination of buspirone and levodopa/carbidopa, and placebo.
  -Participants' muscle activity will be assessed during a 10MWT with EMGs.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Bloch, Pr MD, Principal Investigator — CHUV
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The SAP, CSR, AEs, SAEs will be made available to other researchers once the study is completed and data have been analyzed
Supporting Information: SAP, CSR
Time Frame: Three years after

REFERENCES:
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Formento E, Minassian K, Wagner F, Mignardot JB, Le Goff-Mignardot CG, Rowald A, Bloch J, Micera S, Capogrosso M, Courtine G. Electrical spinal cord stimulation must preserve proprioception to enable locomotion in humans with spinal cord injury. Nat Neurosci. 2018 Dec;21(12):1728-1741. doi: 10.1038/s41593-018-0262-6. Epub 2018 Oct 31. PMID 30382196
- See also: Courtine-Lab is a part of the Center for Neuroprosthetic and Brain Mind Institute of the Life Science School at the Swiss Federal Institute of Technology Lausanne (EPFL). The laboratory is headed by Professor Courtine — http://courtine-lab.epfl.ch/
- See also: The clinical trial is located at the CHUV in Lausanne, Switzerland. — https://www.chuv.ch/fr/chuv-home/